CLINICAL TRIAL: NCT06776536
Title: Evaluation of Rectal Infiltration Depth and Length in Bowel Involvement of Deep Infiltrative Endometriosis (DIE) Using Intraoperative Transrectal Ultrasound (TRUS)
Acronym: DIE IO TRUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Baris KAYA, Associate Professori,MD, Başakşehir Çam & Sakura City Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: E-96317027-514.10-263823748
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Deep Infiltrating Endometriosis (DIE); Transrectal Ultrasound; Bowel Endometriosis; Bowel Resection
Keywords: Deeply infiltrating endometriosis; bowel endometriosis; transrectal ultrasound; bowel resection

STUDY DESIGN:
Masking Description: The radiologist (A) interpreting the preoperative MRI and the radiologist (B) performing the intraoperative TRUS will be different individuals. The radiologist performing the TRUS will be blinded to the patient's clinical information and MRI findings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Evaluation of Rectal Infiltration Depth and Length in Bowel Infiltrating Endometriosis (Experimental): This study aims to investigate the feasibility of measuring the depth and extent of bowel involvement using intraoperative transrectal ultrasound in patients undergoing surgery for intestinal endometriosis
  Interventions: Diagnostic Test: Transrectal ultrasound of the bowel endometriosis during operation

INTERVENTIONS:
Diagnostic Test: Transrectal ultrasound of the bowel endometriosis during operation — This is a prospective, single-arm study aimed at evaluating the efficacy of intraoperative transrectal ultrasound (TRUS) in assessing rectal infiltration depth and length in patients with bowel involvement due to deep infiltrative endometriosis (DIE). The study will include 15-40 female patients aged 18-55, diagnosed with intestinal endometriosis preoperatively using transvaginal ultrasound and MRI, and scheduled for bowel resection.
  Preoperative evaluations will include pelvic examination, imaging (TVUS and MRI), and pain assessment using a visual analog scale (VAS). During surgery, TRUS will be used to measure the depth and length of rectal involvement, and findings will be compared with preoperative MRI results.

SUMMARY:
we aim to evaluate the success of intraoperative transrectal ultrasound in measuring the depth and extent of bowel involvement in patients preoperatively diagnosed with intestinal endometriosis using transvaginal ultrasound and MRI, and who are planned for bowel resection

DETAILED DESCRIPTION:
This is a prospective, single-arm study aimed at evaluating the efficacy of intraoperative transrectal ultrasound (TRUS) in assessing rectal infiltration depth and length in patients with bowel involvement due to deep infiltrative endometriosis (DIE). The study will include 15-40 female patients aged 18-55, diagnosed with intestinal endometriosis preoperatively using transvaginal ultrasound and MRI, and scheduled for bowel resection.

Preoperative evaluations will include pelvic examination, imaging (TVUS and MRI), and pain assessment using a visual analog scale (VAS). During surgery, TRUS will be used to measure the depth and length of rectal involvement, and findings will be compared with preoperative MRI results. Data will be analyzed using statistical methods, including sensitivity, specificity, and ROC curve analysis, to determine the diagnostic performance of TRUS.

The study will be conducted at Istanbul Başakşehir Çam and Sakura City Hospital, with multidisciplinary contributions from gynecology, radiology, and general surgery teams.

ELIGIBILITY:
Inclusion Criteria:

* The study will include a minimum of 15 female patients aged 18-55 with bowel involvement due to deep infiltrative endometriosis, requiring bowel resection.

Exclusion Criteria:

Patients with bowel endometriosis who does not require bowel resection, patients who have other bowel diseases, such as rectal tumors, Crohn's disease, or ulcerative colitis, will be excluded.

-

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female with deep endometriosis patients with bowel endometriosis will be enrolled
Enrollment: 15 (Estimated)
Dates: Start 2025-01-07 (Estimated); Primary Completion 2026-04-07 (Estimated); Study Completion 2026-04-07 (Estimated)

PRIMARY OUTCOMES:
Intraoperative transrectal ultrasound of the rectal involvement of the deep infiltrating endometriosis will be compared with preoperative MRI | From enrollment to the 16 months
  Patients diagnosed with rectal endometriosis and planned for bowel resection will undergo intraoperative transrectal ultrasound during laparoscopy. The transrectal ultrasound will be performed by a blinded radiologist, and the location, depth, and length of rectal involvement in DIE will be measured in millimeters using TRUS. These findings will be recorded. The results will be compared with preoperative MRI results which was performed by another radiologist for this study.

SECONDARY OUTCOMES:
Demographic informations, patient characteristics, disease related pain scores, surgical informations | From enrollment to 16 months.
  Patient demographic information, including age, BMI, known comorbidities, mode and number of deliveries, previous surgeries, and preoperative medical treatments, will be collected. Pain characteristics and visual analog score (VAS) scores for dysmenorrhea, dyspareunia, dysuria, dyschezia, and chronic pelvic pain will be retrieved from the hospital records or patient files. Surgical parameters, such as the type and duration of surgery will be recorded. Early postoperative complications will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Baris Kaya, Associate Professor,MD, Principal Investigator — Başakşehir Çam & Sakura City Hospital
Locations (1):
- Basaksehir Cam ve Sakura City Hospital, Başakşehir Mahallesi G-434 Caddesi No: 2L Başakşehir / İSTANBUL, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
"IPD will not be shared due to concerns regarding patient confidentiality and privacy, as well as the sensitivity of the data related to rectal endometriosis and intraoperative findings.

REFERENCES:
- [Background] Hardman D, Bennett R, Mikhail E. Laparoscopic shaving of rectosigmoid deep infiltrating endometriosis under laparoscopic ultrasound guidance. Fertil Steril. 2023 Jul;120(1):206-207. doi: 10.1016/j.fertnstert.2023.04.026. Epub 2023 Apr 26. PMID 37116640
- [Background] Hudelist G, Ballard K, English J, Wright J, Banerjee S, Mastoroudes H, Thomas A, Singer CF, Keckstein J. Transvaginal sonography vs. clinical examination in the preoperative diagnosis of deep infiltrating endometriosis. Ultrasound Obstet Gynecol. 2011 Apr;37(4):480-7. doi: 10.1002/uog.8935. PMID 21433168
- [Background] Griffiths A, Koutsouridou R, Vaughan S, Penketh R, Roberts SA, Torkington J. Transrectal ultrasound and the diagnosis of rectovaginal endometriosis: a prospective observational study. Acta Obstet Gynecol Scand. 2008;87(4):445-8. doi: 10.1080/00016340801948318. PMID 18382872
- [Background] Doniec JM, Kahlke V, Peetz F, Schniewind B, Mundhenke C, Lohnert MS, Kremer B. Rectal endometriosis: high sensitivity and specificity of endorectal ultrasound with an impact for the operative management. Dis Colon Rectum. 2003 Dec;46(12):1667-73. doi: 10.1007/BF02660773. PMID 14668593
- [Background] Roman H, Kouteich K, Gromez A, Hochain P, Resch B, Marpeau L. Endorectal ultrasound accuracy in the diagnosis of rectal endometriosis infiltration depth. Fertil Steril. 2008 Oct;90(4):1008-13. doi: 10.1016/j.fertnstert.2007.07.1361. Epub 2007 Nov 26. PMID 18023444
- See also: The European Endometriosis League (EEL) h The aim is to extend public awareness and support scientific research in the field of Endometriosis — https://euroendometriosis.com/
- Available data/document: institutional review board — https://camsakurasehir.saglik.gov.tr/